CLINICAL TRIAL: NCT07371936
Title: Analysis of Pediatric Trauma Registry Data:Patterns,Outcomes, and Predictors of Injury Severity.
Brief Title: Analysis of Pediatric Trauma Registry Data:Patterns,Outcomes,and Predictors of Injury Severity.
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, Maria Wageh Youssef Fahem, Resident at Emergency Medicine Department, Sohag University
Other Study IDs: Soh-Med--25-12-12MS
Record Dates: First submitted 2026-01-01; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Analysis of Pediatric Trauma
Keywords: Pediatric trauma; Patterns; Morbidity; Mortality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Type of the study: A prospective analytical observational study using pediatric trauma registry data.

Study period: The study will last for six months. Study setting: Sohag and Alexandria University Hospitals, Department of Emergency Medicine and pediatric surgery department .

DETAILED DESCRIPTION:
Study subject:

Inclusion criteria:

* Pediatric patients aged less than 18 years.
* Presenting with any form of traumatic injury.

Exclusion Criteria:

* Patients dead on arrival without available prehospital information.
* Non-traumatic medical emergencies recorded in error.
* pediatric patients presenting with burn.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged less than 18 years.
* Presenting with any form of traumatic injury.

Exclusion Criteria:

* Patients dead on arrival without available prehospital information.
* Non-traumatic medical emergencies recorded in error.
* pediatric patients presenting with burn.

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sohag and Alexandria University Hospitals, Department of Emergency Medicine and pediatric surgery department .
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
ICU admission rate. | Six months
  The number and percentage of patients admitted to the intensive care unit during the index hospitalization among all eligible pediatric injury patients.

SECONDARY OUTCOMES:
length of hospital stay | Six months
  Differences in length of hospital stay among injury types.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
I don't decide till now